CLINICAL TRIAL: NCT04853186
Title: Cholera Control in Endemic Regions of Africa: Clinical Surveillance and Cholera Shedding Study in the Context of Mass Vaccination Campaigns, Democratic Republic of the Congo
Brief Title: Impact Study of Cholera Vaccination in Endemic Areas - Clinical Surveillance
Status: Recruiting | Type: Observational
Sponsor: Epicentre (Other)
Collaborators: Wellcome Trust (Other); Médecins Sans Frontières, France (Other); Ministry of Public Health, Democratic Republic of the Congo (Other Government); Institut National de Recherche Biomédicale. Goma, République Démocratique du Congo (Unknown); Grand Labo de Lubumbashi (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2104-WT; 215689/Z/19/Z (Other Grant/Funding Number: Wellcome Trust)
Record Dates: First submitted 2021-04-16; First posted 2021-04-21 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cholera
Keywords: Cholera incidence rates; Mass vaccination campaign; V.Cholerae
MeSH Terms: conditions — Cholera

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fresh stool samples will be systematically collected for patients presenting at the CTC and fulfilling the cholera case definition.Samples will first be tested with rapid test, then humid filter papers (for culture) and dry filter papers (for PCR) will be made from fresh sample.Enriched rapid tests could also be tested if appropriate to enhance RDT specificity.A fresh stool sample will be collected from all household members upon household visits.On day 90and180, fresh stool samples will only be collected from household member having tested positive for active cholera shedding during the course of the previous visits.Samples from peri-household environment including drinking water, kitchen swab, latrine swab and latrins sludge, will be taken during the first three household visits and sent to laboratory for testing.Peri-household environment samples collection will be stopped afterwards upon the course of the follow-up if all of them tested negative for at least2 consecutive visits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This project aims to fill this essential knowledge gap by assessing the impact of oral cholera vaccine mass campaigns in 2 sites (urban and rural) in DRC, described in this protocol. The evidence generated from this project will be key to develop future strategies regarding cholera vaccine use in endemic settings, including places with higher burden in terms of cholera mortality.

DETAILED DESCRIPTION:
The project will comprise three different components:

1. Clinical cholera surveillance to measure cholera diseases incidence in selected African hotspots targeted by vaccination.
2. Serial serological surveys to measure the prevalence of recent cholera infection (within the last 12 months).
3. Identification and follow up of individuals with positive V. cholerae shedding (symptomatic or asymptomatic) among sero-survey participants and among household members of cholera confirmed cases.

The present protocol relates to the setup of clinical surveillance and the follow up of individuals with positive V. cholerae shedding identified through clinical surveillance, in DRC.

This protocol will allow us to assess if a large vaccination campaign reaching high coverage in cholera hotspot in Africa can allow sustained control of cholera for at least two years, by fulfilling the following specific objectives:

* To measure cholera incidence rates following the mass vaccination campaign in two cholera hotspots in Africa.
* To assess the duration of shedding among vaccinated and unvaccinated individuals and the duration of viable V. cholerae in the peri-household environment.
* To measure the secondary cholera attack rates (symptomatic and asymptomatic) at household level among vaccinated and unvaccinated individuals following the identification of an index case in a given household.
* To describe the global genetic diversity of V. cholerae strains in the study areas and within households affected by cholera.
* To develop sustainable surveillance methods that could be applied in other hotspots in Africa and elsewhere aiming to monitor the impact of the cholera control program.

ELIGIBILITY:
For Surveillance in study CTCs

Inclusion Criteria:

* All patients presenting at the time of the study to any selected Cholera Treatment Center/Cholera Treatment Unit (CTC/CTU), matching the case definition and giving his/her consent (or assent for children 8 to 17 years old) to participate in the study will be eligible.

Exclusion Criteria:

* Patients who decline to participate will be excluded from the study.

Follow up of individuals with active cholera shedding:

Inclusion Criteria:

1. present to any selected CTC/CTU, match the case definition, participate to the clinical surveillance activity and test positive to RDT OR
2. Be a household member of a person respecting inclusion criteria 1. AND for whom the head of the household has provided verbal consent to participate AND giving his/her consent (or assent for children 8 to 17 years old) to participate in the study will be eligible.

Exclusion Criteria:

- Individuals who decline to participate will be excluded from the study, as well as households for whom the head of the household (and his or her representative) decline the participation of his/her household.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients presenting to a CTC/UTC with a watery diarrhoea (≥ 3 watery stools per day), with or without vomiting, with or without dehydration.
  For the follow-up of individuals with active cholera shedding:
  This activity will take place in the community at included patient's households. Patients will be identified through CTC/CTUs and will therefore be conducted in the catchment area of these structures.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2021-05-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To better characterize cholera transmission in cholera hotspot in Africa and assess the impact of a large vaccination campaign reaching high coverage on sustained control of cholera transmission for at least two years. | 2 years
  Specific objectives 1 and 4 will be answered through the clinical surveillance activity, below referred to as "Surveillance in study CTCs", while 2 and 3 relate to the follow-up activity, below referred to as "Follow-up of individuals with active cholera shedding".

SECONDARY OUTCOMES:
1. To retrospectively study surveillance data, and prospectively measure cholera incidence rates of medically-attended confirmed cases following the mass vaccination campaign in two cholera hotspots in Africa. | 2 years
2. To assess the duration of shedding among vaccinated and unvaccinated individuals and the duration of viable V. cholerae in the peri-household environment. | one year
3. To measure the secondary cholera attack rates (symptomatic and asymptomatic) at household level among vaccinated and unvaccinated individuals following the identification of an index case in a given household. | one year
4. To describe the global genetic diversity of V. cholerae strains in the study areas and within households affected by cholera. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Klaudia PORTEN, Study Director — Epicentre; Francesco Luquero, Study Chair — GAVI
Locations (1):
- Anais Broban, Goma, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: Undecided
Datasets gathered during this study are susceptible to be made available to other research groups which are currently actively collaborating with Epicentre in the cholera research projects. In that case, data sharing agreements will be made with the relevant research groups.